CLINICAL TRIAL: NCT04383626
Title: Fear and Practice Modification Among Dentists During COVID-19 Pandemic
Brief Title: Fear Among Dentists During COVID-19 Pandemic
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mariam Mohsen Aly, lecturer in pediatric dentistry and dental public health, faculty of dentistry, Cairo university, Cairo University
Other Study IDs: COVID-19 pandemic
Record Dates: First submitted 2020-05-10; First posted 2020-05-12 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: COVID
Keywords: fear; practice modification; COVID-19; epidemic
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aimed to evaluate the anxiety and fear of infection between dentists working during the present corona virus disease 2019 (COVID-19) pandemic and to explore dentist's knowledge about various practice modifications and guidelines to fight the novel corona virus

DETAILED DESCRIPTION:
The spread of corona virus (COVID-19) has posed significant challenges for dentistry and medicine, and dental and medical schools, in all affected countries.

The speed of reaction and type of response to this disease around the world have been very variable according to differing healthcare systems, economies and political ideologies

ELIGIBILITY:
Inclusion Criteria:

* Dentist having bachelor of dentistry or equivalent degree

Exclusion Criteria:

* paramedical staff and dental students

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Dentist having bachelor of dentistry or equivalent degree
Sampling Method: Probability Sample
Enrollment: 216 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2020-04-05 (Actual); Study Completion 2020-05-05 (Actual)

PRIMARY OUTCOMES:
fear among dentist during COVID 19 epidemic | 1 week
  measuring unit questionnaire and the measuring unit is categorical yes, no and unaware

SECONDARY OUTCOMES:
practice modification among dentist during COVID 19 epidemic | 1 week
  measuring unit questionnaire and the measuring unit is categorical yes, no and don't know

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt